CLINICAL TRIAL: NCT00226213
Title: Peripherally Inserted Central Catheter Placement by Interventional Radiologists Using the Sonic Flashlight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0406143
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Catheterization

INTERVENTIONS:
Procedure: Peripherally Inserted Central Catheter Placement

SUMMARY:
The purpose of the study is to perform the first clinical trial on human subjects using the Sonic Flashlight (SF) to guide placement of Peripherally Inserted Central Catheters (PICCs).

DETAILED DESCRIPTION:
The SF prototype is an ultrasound (US) display device under development at our institution that replaces the traditional US monitor by using a half -silvered mirror to reflect real-time US images into the body. When the operator looks through the half -silvered mirror, the US image appears to float beneath the surface of the skin, exactly where it is being scanned. The SF merges the US image, probe, needle, operator's hands, and patient into the same field of view, making procedures more intuitive to the novice user, in contrast to conventional US (CUS) guided procedures, where hand-eye coordination is displaced, forcing the operator to look away from the field to see the US screen. We have previously shown that VA in phantoms is easier to use, faster to use, and faster to learn than CUS in novice and experienced US users. The current SF prototype uses a 10MHz US system (Terason, Burlington, MA) modified by attaching a small flat-panel display (AM550L OLED, Kodak, Rochester, NY) and a 20x50x1mm half -silvered mirror to the probe. A standard, clear, sterile polyethylene US probe cover was placed over the entire SF to sterilize the device. 15 subjects needing PICC lines were enrolled in this study. Scanning the upper arm of each patient with the SF, the basilic vein, brachial vein, and brachial artery were identified on the in situ US image. A 21ga needle was guided into the basilic or brachial vein. The number of attempts, or sticks, per PICC line placement, specific vein accessed, and reason for a failed attempt were recorded.

The vasculature was clearly visualized in situ using the SF. The needle was aimed and easily inserted into the basilic or brachial vein, and the needle tip visualized at its expected location. Successful vascular access was obtained with all 15 subjects, 13 of 15 on the first attempt, and 2 of 15 on the second attempt. 3 of the 15 lines encountered mild blurriness looking through the SF due to inconsistent optical properties of the probe cover.

This study shows that venous access can be obtained using the SF. Once the optical problems with the probe covers are addressed, the SF will be ready for a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing a PICC line insertion as part of their standard care

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
PICC lines successfully placed using the Sonic Flashlight

SECONDARY OUTCOMES:
PICC lines successfully placed using conventional ultrasound machines

CONTACTS AND LOCATIONS:
Overall Officials: George D Stetten, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States